CLINICAL TRIAL: NCT04396938
Title: The Effect of a Single Dose of Lamotrigine on Brain Function in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R49749/RE003
Record Dates: First submitted 2019-09-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lamotrigine (Experimental): Single dose of Lamotrigine (300mg - capsule). In healthy volunteers.
  Interventions: Drug: Lamotrigine
- Placebo (Placebo Comparator): Placebo capsule: identical appearance to experimental capsule. In healthy volunteers.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lamotrigine — Active Drug Capsule
  Arms: Lamotrigine
Drug: Placebos — Placebo Capsule
  Arms: Placebo

SUMMARY:
This study will test whether a single dose of Lamotrigine (300mg) exerts significant effects on emotional processing, cognitive ability and neural activity in healthy volunteers compared to placebo.

DETAILED DESCRIPTION:
Glutamate has been implicated in the aetiology of mood disorders and there is current interest in developing novel agents targeting this system. However, the role of glutamate in human emotional function is relatively unknown. Lamotrigine's pharmacological profile involves a blockade of voltage-gated sodium channels, leading to an inhibition in the release of glutamate and resulting in a general inhibitory effect on cortical neuronal function.

The current study plans to investigate the effects of modifying glutamate on emotional processing, cognitive function and neural activity. For this, 36 healthy volunteers will be recruited to the study and randomised to receive a single dose of lamotrigine (300 mg) or placebo. Two hours after drug administration, the effects of emotional processing via the use of cognitive tasks will be assessed using fMRI. This will be followed by an emotional test battery that will measure aspects of cognitive function as well.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-40 years
* Willing and able to give informed consent for participation in the study
* Sufficiently fluent English to understand and complete the task

Exclusion Criteria:

* Current usage of psychoactive medication
* Current usage of the contraceptive pill
* Any past or current Axis 1 DSM-IV psychiatric disorder
* Significant medical condition
* Current pregnancy or breastfeeding
* Current or past history of drug or alcohol dependency
* Participation in a psychological or medical study involving the use of medication within the last 3 months
* Previous participation in a study using the same, or similar, emotional processing tasks
* Smoker > 5 cigarettes per day
* Typically drinks > 6 caffeinated drinks per day
* Takes folic acid supplements
* History of recurrent allergies and rashes
* Contraindication to MRI (e.g. claustrophobia and metallic implants)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Neural function | Data reporting and analysis to be completed within 1 year following study completion.
  fMRI resting state analysis
Neural function | Data reporting and analysis to be completed within 1 year following study completion.
  fMRI task analysis
Neural function | Data reporting and analysis to be completed within 1 year following study completion.
  fMRI checkerboard analysis

SECONDARY OUTCOMES:
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Analysis of recognition of emotion in faces (an Emotional Test Battery component)
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Speed of negative self-descriptor processing (an Emotional Test Battery component)
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Emotional memory analysis (an Emotional Test Battery component)
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Beck Depression inventory (BDI) questionnaire analysis
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Positive and negative affect schedule (PANAS) questionnaire analysis
Emotional Processing and Cognitive Function | Data reporting and analysis to be completed within 6 months following study completion.
  Stait-trait anxiety inventory (STAI) questionnaire analysis

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calabrese JR, Huffman RF, White RL, Edwards S, Thompson TR, Ascher JA, Monaghan ET, Leadbetter RA. Lamotrigine in the acute treatment of bipolar depression: results of five double-blind, placebo-controlled clinical trials. Bipolar Disord. 2008 Mar;10(2):323-33. doi: 10.1111/j.1399-5618.2007.00500.x. PMID 18271912
- [Background] Deakin JF, Lees J, McKie S, Hallak JE, Williams SR, Dursun SM. Glutamate and the neural basis of the subjective effects of ketamine: a pharmaco-magnetic resonance imaging study. Arch Gen Psychiatry. 2008 Feb;65(2):154-64. doi: 10.1001/archgenpsychiatry.2007.37. PMID 18250253
- [Background] Doyle OM, De Simoni S, Schwarz AJ, Brittain C, O'Daly OG, Williams SC, Mehta MA. Quantifying the attenuation of the ketamine pharmacological magnetic resonance imaging response in humans: a validation using antipsychotic and glutamatergic agents. J Pharmacol Exp Ther. 2013 Apr;345(1):151-60. doi: 10.1124/jpet.112.201665. Epub 2013 Jan 31. PMID 23370794
- [Background] Murphy SE, Norbury R, O'Sullivan U, Cowen PJ, Harmer CJ. Effect of a single dose of citalopram on amygdala response to emotional faces. Br J Psychiatry. 2009 Jun;194(6):535-40. doi: 10.1192/bjp.bp.108.056093. PMID 19478294